CLINICAL TRIAL: NCT02419703
Title: The STAR™ Tumor Ablation Registry
Status: Terminated | Type: Observational
Why Stopped: Difficulty Enrolling
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: DFINE Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DF-15-03
Record Dates: First submitted 2015-04-10; First posted 2015-04-17 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Lesions in Vertebral Bodies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving Targeted Radiofrequency Ablation (t-RFA)
  Interventions: Device: STAR™ Tumor Ablation System

INTERVENTIONS:
Device: STAR™ Tumor Ablation System — Targeted Radiofrequency ablation of painful metastatic tumor in the vertebral body.

SUMMARY:
Registry collecting data on use of The STAR™ Tumor Ablation System.

DETAILED DESCRIPTION:
The STAR Prospective Registry is an observational registry to gather clinical safety and outcome data in patients with painful spinal metastases in the thoracolumbar spine (T1-L5) following targeted radiofrequency ablation (t-RFA) treatment with the STAR™ Tumor Ablation System.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with painful spinal metastatic lesions in thoracolumbar vertebrae (T1-L5) that will be treated with t-RFA using the STAR™ Tumor Ablation System.
* Have signed informed consent

Exclusion Criteria:

* Subjects under 18 years old
* Subjects with heart pacemakers, or other electronic device implants
* Subjects intended for t-RFA in vertebral body levels C1-7

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with painful spinal metastatic lesions in thoracolumbar vertebrae (T1-L5) that will be treated with t-RFA using the STAR™ Tumor Ablation System.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

PRIMARY OUTCOMES:
Pain relief (Numerical Rating Pain Scale), post t-RFA | 1 month
  measured by Numerical Rating Pain Scale (NRPS, 0-10 scale)

SECONDARY OUTCOMES:
Pain & Quality of Life Improvement (measured by the FACT G7 & Numerical Rating Pain Scale) | 1 week, 1 month, 3 month, 6 month, 12 month
  measured by the FACT G7 & Numerical Rating Pain Scale

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - John Muir Medical Center, Concord, California
  - Southern California Institute of Neurological Surgery, Escondido, California
  - University of California, Los Angeles, Los Angeles, California
  - St. Joseph's Medical Center, Stockton, California
  - University of Colorado, Denver, Colorado
  - Mori Bean and Brook Radiology, Jacksonville, Florida
  - Medical Imaging & Therapeutics, Lady Lake, Florida
  - VIR Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - University of Tennessee, Knoxville, Tennessee
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin